CLINICAL TRIAL: NCT03282890
Title: Testing an Integrated Bio-Behavioral Primary HIV Prevention Intervention Among High-Risk People Who Use Drugs
Acronym: CHRP-BB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); APT Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Michael Copenhaver, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H17-200; R01DA044867 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Risk Behavior; HIV/AIDS; Medication Adherence; Substance Abuse
Keywords: HIV; Substance Abuse; Pre-Exposure Prophylaxis; HIV Risk Behavior; Methadone Maintenance
MeSH Terms: conditions — Risk-Taking; Acquired Immunodeficiency Syndrome; Medication Adherence; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHRP-BB (Experimental): Patients assigned to the CHRP-BB will receive a weekly HIV risk reduction and PrEP adherence group level intervention led by two facilitators trained and supervised by the PI, a licensed clinical psychologist. It is a substantially shortened version of the comprehensive Holistic Health Recovery Program (HHRP)-based interventions that have been identified as demonstrating evidence of effectiveness in two randomized clinical trials. The CHRP-BB, which includes four 50-minute groups (1 group per week), will contain only content that relates explicitly to drug- or sex-related HIV risk reduction and PrEP adherence. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).
  Interventions: Other: CHRP-BB
- Control Condition (No Intervention): The time-and-attention-matched control condition for the proposed research will be a time and contact-matched, non-contaminating support group for individuals in recovery modeled after similar groups offered in the community. There will be no overlap between the content of the comparison intervention and experimental intervention although the basic structure will be the same. Thus, each participant will be asked to attend four 50-minute weekly group sessions led by two trained facilitators. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).

INTERVENTIONS:
Other: CHRP-BB — The CHRP-BB intervention is a theory-based, manual-guided, HIV risk reduction and PrEP adherence intervention. It is an integrated evidence-based intervention that uses a coping skills training approach to primary prevention and is delivered in a small group modality by two trained intervention facilitators using a motivational enhancement therapeutic style to address high risk drug- and sex-related HIV risk behaviors and PrEP adherence. Importantly, the CHRP-BB intervention includes specific behavioral and mHealth strategies designed and tested to accommodate difficulties stemming from moderate to severe neuro-cognitive impairment (NCI).
  Arms: CHRP-BB

SUMMARY:
This study will evaluate the efficacy and cost-effectiveness of CHRP-BB - an integrated bio-behavioral approach that incorporates the use of PrEP - with an evidence-based behavioral approach aimed at enhancing PrEP adherence and HIV risk reduction among high risk PWUD.

DETAILED DESCRIPTION:
PWUD remain a priority population as they represent a critical conduit for new HIV infections, which are transmitted through preventable drug- and sex-related HIV risk behaviors. Pre-Exposure Prophylaxis (PrEP) - the daily self-administration of antiretroviral medication - has enormous potential to bolster primary HIV prevention outcomes among PWUD. PrEP is a FDA-approved biomedical HIV prevention strategy recommended by the CDC and WHO for key populations, including PWUD. Despite unequivocal evidence supporting PrEP, its scale-up has been nearly absent among high risk PWUD. Moreover, adherence to PrEP is crucial if it is to be effective with high risk individuals. Recent research, however, indicates that optimal PrEP adherence may be compromised by neurocognitive impairment (NCI), particularly among PWUD. Due to chronic drug use, related lifestyle experiences, and other health challenges, many PWUD experience NCI to the extent that it impedes medication adherence, HIV risk reduction, and treatment retention. In a recent HIV prevention trial, over a third of high risk PWUD on opioid replacement therapy (ORT) had moderate to high levels of NCI and, moreover, were less likely to reduce their HIV transmission risk vs. those without NCI. The potentially disruptive impact of NCI must therefore be addressed when designing contemporary intervention strategies targeting PWUD. Contemporary approaches must also be cost-effective and usable in real-world treatment settings, such as methadone maintenance programs (MMPs) where high risk PWUD are concentrated and can be readily reached with primary prevention. To date, however, primary prevention efforts have largely relied on singular strategies (e.g., methadone or PrEP alone) with modest HIV risk reduction outcomes for PWUD. Instead, advancing combination approaches capable of harnessing the synergy and efficiency possible via multiple evidence-based strategies is most effective. This combination strategy is especially important when intervening with high risk PWUD with NCI due to the potential decreased effectiveness of PrEP when adherence is suboptimal, thereby necessitating behavioral interventions that focus on reducing HIV risk and increasing PrEP adherence. Building on promising preliminary work, the proposed trial will fill a critical void by testing an integrated bio-behavioral approach that incorporates the use of PrEP with an evidence-based behavioral approach and, using innovative strategies, enhances PrEP adherence and HIV risk behavior in a manner that accommodates NCI among PWUD.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-V criteria for opioid-dependence and are enrolled in methadone maintenance drug treatment at the APT Foundation, Inc.
* Were confirmed to be HIV-negative and started on PrEP in the past week
* Report unsafe injection drug use practices or unprotected sex within the past 3 months
* Have a cell phone
* Are able to read and understand the questionnaires, ACASI, and informed consent form
* Available for the full duration of the study with no anticipated circumstances impeding participation (e.g., pending charges, jail term).

Exclusion Criteria:

* Have an untreated bipolar or psychotic disorder
* Are actively suicidal or homicidal as assessed by trained research staff under the supervision of a licensed clinical psychologist
* Cannot speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Copenhaver, PhD, Principal Investigator — University of Connecticut
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shrestha R, Altice F, Karki P, Copenhaver M. Developing an Integrated, Brief Biobehavioral HIV Prevention Intervention for High-Risk Drug Users in Treatment: The Process and Outcome of Formative Research. Front Immunol. 2017 May 11;8:561. doi: 10.3389/fimmu.2017.00561. eCollection 2017. PMID 28553295
- [Background] Shrestha R, Karki P, Altice FL, Huedo-Medina TB, Meyer JP, Madden L, Copenhaver M. Correlates of willingness to initiate pre-exposure prophylaxis and anticipation of practicing safer drug- and sex-related behaviors among high-risk drug users on methadone treatment. Drug Alcohol Depend. 2017 Apr 1;173:107-116. doi: 10.1016/j.drugalcdep.2016.12.023. Epub 2017 Feb 2. PMID 28214391
- [Background] Huedo-Medina TB, Shrestha R, Copenhaver M. Modeling a Theory-Based Approach to Examine the Influence of Neurocognitive Impairment on HIV Risk Reduction Behaviors Among Drug Users in Treatment. AIDS Behav. 2016 Aug;20(8):1646-57. doi: 10.1007/s10461-016-1394-x. PMID 27052845
- [Background] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Background] Shrestha R, Huedo-Medina TB, Altice FL, Krishnan A, Copenhaver M. Examining the Acceptability of mHealth Technology in HIV Prevention Among High-Risk Drug Users in Treatment. AIDS Behav. 2017 Nov;21(11):3100-3110. doi: 10.1007/s10461-016-1637-x. PMID 28025735
- [Background] Copenhaver MM, Lee IC, Margolin A. Successfully integrating an HIV risk reduction intervention into a community-based substance abuse treatment program. Am J Drug Alcohol Abuse. 2007;33(1):109-20. doi: 10.1080/00952990601087463. PMID 17366251
- [Background] Copenhaver MM, Lee IC, Baldwin P. A randomized controlled trial of the community-friendly health recovery program (CHRP) among high-risk drug users in treatment. AIDS Behav. 2013 Nov;17(9):2902-13. doi: 10.1007/s10461-013-0539-4. PMID 23835735
- [Background] Avants SK, Margolin A, Usubiaga MH, Doebrick C. Targeting HIV-related outcomes with intravenous drug users maintained on methadone: a randomized clinical trial of a harm reduction group therapy. J Subst Abuse Treat. 2004 Mar;26(2):67-78. doi: 10.1016/S0740-5472(03)00159-4. PMID 15050083
- [Background] Shrestha R, Karki P, Altice FL, Dubov O, Fraenkel L, Huedo-Medina T, Copenhaver M. Measuring Acceptability and Preferences for Implementation of Pre-Exposure Prophylaxis (PrEP) Using Conjoint Analysis: An Application to Primary HIV Prevention Among High Risk Drug Users. AIDS Behav. 2018 Apr;22(4):1228-1238. doi: 10.1007/s10461-017-1851-1. PMID 28695388
- [Background] Shrestha R, Karki P, Huedo-Medina TB, Copenhaver M. Intent to Use Preexposure Prophylaxis (PrEP), HIV Risk Behaviors, and Self-Report Neurocognitive Symptoms by High-Risk Drug Users: A Mediation Analysis. J Assoc Nurses AIDS Care. 2017 Jul-Aug;28(4):612-621. doi: 10.1016/j.jana.2017.04.005. Epub 2017 Apr 19. PMID 28478870
- [Background] Shrestha R, Altice FL, Huedo-Medina TB, Karki P, Copenhaver M. Willingness to Use Pre-Exposure Prophylaxis (PrEP): An Empirical Test of the Information-Motivation-Behavioral Skills (IMB) Model among High-Risk Drug Users in Treatment. AIDS Behav. 2017 May;21(5):1299-1308. doi: 10.1007/s10461-016-1650-0. PMID 27990587
- See also: University of Connecticut Institute for Collaboration on Health, Intervention, and Policy (InCHIP) — http://chip.uconn.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- CHRP-BB (Experimental Condition): Community-friendly health recovery program - bio-behavioral
- Active Control Condition: Treatment as usual - active control group condition
Period: Overall Study
Arm/Group | CHRP-BB (Experimental Condition) | Active Control Condition
Started | 120 (baseline assessment) | 117 (baseline assessment)
Post-test | 105 | 104
3-month Follow-up | 102 | 101
6-month Follooup | 74 | 75
9-month Follow-up | 68 | 64
Completed | 68 (9-month follow-up completion date) | 64 (9-month follow-up completion date)
Not Completed | 52 | 53

BASELINE CHARACTERISTICS:
Groups:
- CHRP-BB: Community-friendly health recovery program - bio-behavioral
- Active Control Condition: Treatment as usual group condition
- Total: Total of all reporting groups
Arm/Group | CHRP-BB | Active Control Condition | Total
Number analyzed (Participants) | 120 | 117 | 237
Age, Categorical [Count of Participants; unit: Participants] — Frequency of age (categorical)
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 120 | 117 | 237
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] — Age in years
  years | 44 [19 to 64] | 44 [19 to 64] | 44 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 58 | 56 | 114
  Gender: Male | 62 | 61 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 13 | 36
  Not Hispanic or Latino | 96 | 97 | 193
  Unknown or Not Reported | 1 | 7 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 29 | 49
  White | 76 | 68 | 144
  More than one race | 23 | 13 | 36
  Unknown or Not Reported | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  United States | 120 | 117 | 237
Currently unemployed [Number; unit: Participants] | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Pre-exposure Prophylaxis (PrEP) Adherence Behavior
Description: The Pre-exposure prophylaxis (PrEP) adherence behavior scale is an 11-item categorical self-report measure designed to assess how confident a participant is about properly taking their PrEP medication (e.g., "How confident are you that you could make PrEP part of your daily routine?"). The scale requires participants to respond to each of the 11 items about adherence by selecting whether they are either 'Not at all confident', 'Somewhat confident', 'Moderately confident', 'Very confident', or 'Completely confident' about the behavior. The 11 items are summed to create a total score, with higher scores indicating a better PrEP adherence behavior outcome. The possible range of total scores is 0-44.
Time Frame: This is measured immediately post-intervention, and then at 3-months, 6-months, and 9 months post-intervention. Results are reported in the table at 9-months.
Measure: Mean (95% Confidence Interval); unit: score
Groups:
- CHRP-BB (Experimental Condition): community-friendly health recovery program - bio-behavioral (CHRP-BB)
- Active Control Condition: time and attention matched control condition
Arm/Group | CHRP-BB (Experimental Condition) | Active Control Condition
Number analyzed (Participants) | 120 | 117
score | 25.9 [20.4 to 31.3] | 22.8 [18.9 to 26.7]

2. Secondary Outcome: HIV Risk Reduction Behavior
Description: HIV risk reduction behavior was assessed using a 4-item categorical self-report measure designed to assess the participant's self-efficacy about engaging in behaviors to reduce their HIV risk (e.g., 'How hard would it be for you to always use condoms or latex protection if you have oral, vaginal, or anal sex?"). The measure requires participants to select one of five possible responses for each of the four items, indicating whether a behavior would be either 'Very hard to do', 'Fairly hard to do', 'Neither hard nor easy to do', 'Somewhat easy to do', or 'Very easy to do'. Responses to the four items were summed and reversed to create a total score, with higher scores indicating a better HIV risk reduction outcome.The possible range of total HIV risk reduction behavior scores is 4 to 20.
Time Frame: This was assessed immediately post-intervention, and then at 3-months, 6-months, and 9 months post-intervention. Results are reported in the table at 9-months.
Measure: Mean (95% Confidence Interval); unit: score
Arm/Group | CHRP-BB (Experimental Condition) | Active Control Condition
Number analyzed (Participants) | 120 | 117
score | 17.5 [16.8 to 18.1] | 16.2 [15.3 to 17.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each participant at baseline, immediately following the 8-week intervention period, and then 3m, 6m, and 9-months post intervention. The adverse event time frame was 11/20/2017 - 10/13/2023.
Arm/Group | CHRP-BB | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/117
Other Adverse Events (participants affected / at risk) | 0/120 | 0/117

LIMITATIONS AND CAVEATS:
This study examines an innovative approach, as the first PrEP-focused intervention tailored to the cognitive profiles of individuals on MOUD, but there are some limitations worth mentioning. This study only recruited participants who could understand, speak, and read the English language, and participants who had a phone for communicating daily text messages in English. Future studies should measure cognitive functioning more frequently in order to improve the precision of this measurement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03282890/Prot_SAP_000.pdf